CLINICAL TRIAL: NCT02891993
Title: Pilot Study of a Symptom Monitoring Intervention for Hospitalized Patients With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Ryan Nipp, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 16-228
Record Dates: First submitted 2016-08-27; First posted 2016-09-08 (Estimated); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Cancer
Keywords: Cancer Care
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IMPROVED Intervention (Experimental): * Patients randomized to IMPROVED will self-report their symptoms each day using a tablet computer.
  * The clinical team will view reports detailing their patients' symptom burden
  * Clinicians will be provided with a graphic depiction of their patients' daily symptom trajectory for that admission
  Interventions: Other: IMPROVED
- Usual Care (Active Comparator): * Patients randomized to Usual Care will self-report their symptoms each day using a tablet computer
  * Patients will report their symptoms to their clinicians as they usually would
  * Clinicians will not be provided with a graphic depiction of their patients' daily symptom trajectory for that admission
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: IMPROVED — The electronic symptom monitoring intervention, "Improving Management of Patient-Reported Outcomes Via Electronic Data (IMPROVED)," consists of patients self-reporting their symptoms each day using a tablet computer. At morning rounds each day, the clinical team will view reports detailing their patients' symptom burden.
  Arms: IMPROVED Intervention
Other: Usual Care — Participants receiving usual care will also self-report their symptoms each day using tablet computers. However, these patients' clinicians will not receive their symptom reports. Patients randomized to usual care will report their symptoms to their clinicians as they usually would, at their own discretion.
  Arms: Usual Care

SUMMARY:
The purpose of this research study is to address the challenge of symptom management for hospitalized patients with cancer.

DETAILED DESCRIPTION:
Patients with cancer may experience a considerable symptom burden, often requiring hospitalizations for symptom management. This study will pilot test an electronic symptom monitoring intervention, "Improving Management of Patient-Reported Outcomes Via Electronic Data (IMPROVED)," versus usual care in hospitalized patients with cancer.

The goal of this study is test a model where patients' symptoms are monitored during their hospital admission electronically via tablet computers. The investigators are studying whether patients whose clinicians receive their patients' detailed symptom reports each day have improved symptom management compared to those whose clinicians do not receive their patients' detailed symptom reports each day.

The study takes place at Massachusetts General Hospital and involves participating in a study for as long as the participants are admitted to the hospital. The information the investigators collect will help them determine if electronic symptom monitoring improves the care of patients with cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Diagnosed with incurable cancer (defined as receiving treatment with palliative intent as per chemotherapy order entry designation, trial consent forms, or not receiving chemotherapy but followed for incurable disease as per oncology clinic notes)
* Admitted to Lunder at Massachusetts General Hospital
* Verbal fluency in English

Exclusion Criteria:

* Unwilling or unable to participate in the study
* Admitted electively
* Participated during a previous admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2016-09; Primary Completion 2017-06-23 (Actual); Study Completion 2017-12-14 (Actual)

PRIMARY OUTCOMES:
Rates of participant completion of >2 symptom reports | 2 years
  To determine rates of participant completion of >2 symptom reports, the investigators will assess the proportion of enrolled participants who complete of >2 symptom reports.

SECONDARY OUTCOMES:
Rates Of Clinicians Noting Their Patients' Symptom Reports | 2 years
  To determine rates of clinicians noting the symptom reports, the investigators will assess the proportion of clinicians who note their patients' symptom reports.
Rates Of Clinicians Developing An Action Plan In Response To Their Patients' Symptom Reports | 2 years
  To determine rates of clinicians developing an action plan in response to the symptom reports, the investigators will assess the proportion of clinicians who develop an action plan in response to their patients' symptom reports.
Rates Of Clinicians Discussing Their Patients' Symptom Reports | 2 years
  To determine rates of clinicians discussing the symptom reports, the investigators will assess the proportion of clinicians who discuss their patients' symptom reports.
Change In Patients' Symptom Scores | 2 years
  The investigators will compare change in patients' symptom scores from baseline to discharge (using the Edmonton Symptom Assessment System [ESAS] symptom scores measured continuously) between study arms.
Change In Patients' Psychological Distress | 2 years
  The investigators will compare change in patients' psychological distress from baseline to discharge (using the Patient Health Questionnaire-4 [PHQ-4] measured continuously) between study arms.
Change In Patients' Depression Scores | 2 years
  The investigators will compare change in patients' depression scores from baseline to discharge (using the depression questions from the Patient Health Questionnaire-4 [PHQ-4] measured continuously) between study arms.
Change In Patients' Anxiety Scores | 2 years
  The investigators will compare change in patients' anxiety scores from baseline to discharge (using the anxiety questions from the Patient Health Questionnaire-4 [PHQ-4] measured continuously) between study arms.
Rates Of Moderate/Severe Symptoms | 2 years
  The investigators will compare rates of moderate/severe symptoms (defined as ESAS scores ≥4) for each day of hospital admission between study arms.
Rates Of Depression Symptoms | 2 years
  The investigators will compare rates of depression symptoms (defined as a score of 3 or greater on the depression subscale of the PHQ-4) for each day of hospital admission between study arms.
Rates Of Anxiety Symptoms | 2 years
  The investigators will compare rates of anxiety symptoms (defined as a score of 3 or greater on the anxiety subscale of the PHQ-4) for each day of hospital admission between study arms.
Rates Of Moderate/Severe Psychological Symptoms | 2 years
  The investigators will compare rates of psychological symptoms (defined as a score of 6 or greater on the PHQ-4) for each day of hospital admission between study arms.
Rates Of Patient Satisfaction | 2 years
  The investigators will compare rates of patient satisfaction (defined as patients reporting 'very satisfied' using the FAMCARE) for each day of hospital admission between study arms.
Hospital Length Of Stay | 2 years
  The investigators will compare hospital length of stay (measured continuously as days admitted to the hospital) between study arms.
30-Day Readmissions Rates | 2 years
  The investigators will compare 30-day readmissions rates (defined as a hospital readmission within 30 days of prior hospital discharge) between study arms.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Nipp, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts general Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nipp RD, El-Jawahri A, Ruddy M, Fuh C, Temel B, D'Arpino SM, Cashavelly BJ, Jackson VA, Ryan DP, Hochberg EP, Greer JA, Temel JS. Pilot randomized trial of an electronic symptom monitoring intervention for hospitalized patients with cancer. Ann Oncol. 2019 Feb 1;30(2):274-280. doi: 10.1093/annonc/mdy488. PMID 30395144